CLINICAL TRIAL: NCT01731470
Title: Intravesical Liposomes for Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-024
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Interstitial Cystitis; Pelvic Pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain | interventions — Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposomes (Experimental): Liposomes
  Interventions: Biological: Liposomes

INTERVENTIONS:
Biological: Liposomes — Intravesical instillation of liposomes.

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is a poorly understood chronic disorder of unknown etiology consisting of irritative bladder symptoms and pelvic pain that dramatically affects quality of life.

Preclinical study data (obtained by using an IC/PBS model in Sprague-Dawley female rats) have demonstrated normalization of urinary frequency indicating that LP may be a potent protectant of the bladder mucosa against inflammation and irritation. Intravesical LP has so far demonstrated an excellent safety profile and minimal toxicity at concentrations of 2 mg/ml. Thus, we hypothesize that intravesical instillation of LP may form a molecular film on bladder ulcer surfaces in patients with IC and provide a safe, effective, and minimally invasive treatment option to alleviating symptoms.

DETAILED DESCRIPTION:
Liposomes (LP), the treatment article in this proposal, were discovered in the process of exploring a "control" compound when measuring the efficacy of liposomally encapsulated capsaicin for the intravesical treatment of interstitial cystitis. Liposomes are lipid vesicles composed of concentric phospholipid bilayers, which enclose an aqueous interior. Liposomes have the ability to form a molecular film on cell and tissue surfaces and are currently being tested as possible therapeutic agents to promote wound healing. Application of liposomes at the wound surface provides a moist protective film over the wound and augments wound healing without chronic inflammatory reactions in the neodermal layer.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent has been obtained

  * Males and females, at least 18 years of age
  * History of IC/PBS for at least 6 months documented in the medical record
  * Recurring IC/PBS symptoms
  * An average of 8 or more urine voids over a 3-day period, confirmed by the baseline voiding diary
  * Bladder pain score > 4 in the last 24 hours (assessed at screening visit)
  * Previous use of medications and/or treatment(s) for symptom relief
  * Females of child-bearing capability agree to use a reliable form of birth control (condoms and/or oral contraceptives (birth control pills)) during the 4 week course of therapy and 1 week thereafter
  * Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the voiding diaries and self-administered questionnaires

Exclusion Criteria:

* • Subjects currently taking prescribed medications for IC/PBS will be able to continue the medications throughout the course of the study. If the patient cannot be maintained on a stable dose of the medication(s) throughout the treatment and follow-up period they will be excluded.

  * Subjects must not have had intravesical treatment(s)/bladder installations of the following medications: dimethylsulfoxide (DMSO), lidocaine and/or heparin within 1 month prior to study visit 1
  * Pregnant or lactating
  * History of bleeding diathesis
  * Currently on anticoagulant therapy (e.g. warfarin, clopidogrel)
  * Active bleeding peptic ulcer disease
  * Obvious neurological impairment which may be affecting bladder function
  * Known allergy to liposomes and/or egg yolk
  * Current or previous participation in another therapeutic or device study within 6 months of the screening visit
  * The presence of any clinically significant systemic disease or condition that in the opinion of the investigator would make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Peters KM, Hasenau D, Killinger KA, Chancellor MB, Anthony M, Kaufman J. Liposomal bladder instillations for IC/BPS: an open-label clinical evaluation. Int Urol Nephrol. 2014 Dec;46(12):2291-5. doi: 10.1007/s11255-014-0828-5. Epub 2014 Sep 11. PMID 25209396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomes
Started | 16 (Number of patients consented to participate in the study)
Completed | 14 (Number of patients enrolled in the study)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Did not meet study criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Liposomes
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Severity at 4 and 8 Weeks Post-Treatment as Measured by the Total O'Leary-Sant IC Symptom and Problem Index (ICSI/ICPI) Score
Description: The O'Leary-Sant IC Symptom Index (ICS-I) total score ranges from 0 to 20 and the Problem Index (ICP-I) total score ranges from 0 to 16. Each index has 4 questions and lower scores represent a better outcome. A total ICSI/ICPI score is obtained by adding the total scores from both indices. The combined ICSI/ICPI total score ranges from 0 to 36.
Time Frame: 4 and 8 weeks post-treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Liposomes
Number analyzed (Participants) | 14
units on a scale
  Baseline to 4 Weeks Post Treatment | -4 [-7 to -1]
  Baseline to 8 Weeks Post Treatment | -4 [-8 to -1]

2. Secondary Outcome: Change in Pain Scores at 4 and 8 Weeks Post-Treatment as Measured by the Visual Analog Scale (VAS)
Description: Patients utilized the Visual Analog Scale (VAS) to describe their pain. The scale ranges from 0:No pain to 10: Pain as bad as it could possibly be.
Time Frame: 4 and 8 weeks post-treatment
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Liposomes
Number analyzed (Participants) | 14
units on a scale
  Baseline to 4 Weeks Post | -2 [-3.82 to 0.00]
  Baseline to 8 Weeks Post-Treatment | -1.14 [-3.90 to -0.90]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 12 weeks, from the first treatment visit through 8 weeks post-treatment.
Arm/Group | Liposomes
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomes (N=14)
Hematuria (Renal and urinary disorders) | 1 (1)
Irritable Bowel (Gastrointestinal disorders) | 1 (1)
Muscle Pull (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Renal and urinary disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pinched Nerve (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open-label trial without evaluation of placebo effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No